CLINICAL TRIAL: NCT06842667
Title: Development and Preliminary Testing of a "Papageno"-Story Interview Intervention- Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Foundation for Suicide Prevention (Other); Ouida Scholar Award (Unknown)
Responsible Party: Principal Investigator, Jane Harness, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00266531; SRG-1-123-19 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papageno video (Experimental): The arm will watch a compilation of interviews on proximal risk factors for suicide
  Interventions: Behavioral: Papageno video
- Control video (Active Comparator): The arm will watch an educational control video
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Papageno video — The intervention will be a video (14 min 13 sec in length) of a series of clips from the "Papageno" interviews developed during the pilot phase of this project. The decision to combine the videos and shorten the total length of the video was based on the feedback we received during the acceptability and feasibility phase of this study. Interviewees were asked questions about a time in their life when they came close to suicide but found non-suicide alternatives (their "Papageno" story).
  Arms: Papageno video
Behavioral: Control video — The control condition will involve viewing a mental health education video (12 min 14 sec in length) created by our team. It is a simple informational video, aimed at psychoeducation about suicide and safety promotion. It includes a list of mental health and crisis resources. Both videos are interview-style.
  Arms: Control video

SUMMARY:
The purpose of this study is to determine the effects of a short "Papageno story" video of a compilation of interviews on proximal risk factors for suicide. The researchers believe that the intervention may increase protective factors related to suicide.

ELIGIBILITY:
Inclusion Criteria:

* People who are part of an existing cohort within DesignXM
* They will also answer yes to the question: "In the past 1 year, have you wished you were dead or wished you could go to sleep and not wake up?"

Exclusion Criteria:

* No exclusions if all inclusion criteria is met

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 506 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Suicidal ideation | Immediately before and after watching the video and at 3 months
  Assessed with the Abbreviated Reasons For Living- Young Adult Abbreviated (RFL-YA-II) which consists of 24 questions rated on a scale of 1-6. Higher scores indicate greater importance.
Hopelessness | Immediately before and after watching the video and at 3 months
  Assessed with the Beck Hopelessness Scale-4 (BHS-4). The BHS-4 assesses participants' sense of hopelessness, including perceptions of whether their personal actions can improve future outcomes. Participants rate 4 items using a 4 point Likert scale (e.g. "My future seems dark to me"). Each question is coded 0 for positive expectations and 1 for negative expectations.

SECONDARY OUTCOMES:
Participant perceived agency | Immediately before and after watching the video and at 3 months
  As measured by the Perceived Control Scale which is a single-item measure of participant perceived control. Participants will rate agreement with the statement, "right now, I feel like things are out of my control" from 0-10 ("not at all" to "a lot").

CONTACTS AND LOCATIONS:
Overall Officials: Jane Harness, DO, Principal Investigator — University of Michigan; Cheryl King, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported.
Supporting Information: Study Protocol
Time Frame: Approximately 5 years following publication.
Access Criteria: Investigators whose proposed use of the data has been approved by the investigator.